CLINICAL TRIAL: NCT06318598
Title: Dissezione Fenotipica Guidata da Biomarcatori Della Sclerosi Laterale Amiotrofica/Biomarker-driven Phenotypic Dissection of Amyotrophic Lateral Sclerosis
Brief Title: Biomarker-driven Phenotypic Dissection of Amyotrophic Lateral Sclerosis
Acronym: DRIVEALS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other); Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: 23M202
Record Dates: First submitted 2024-03-08; First posted 2024-03-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma, serum, CSF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to understand the clinical variability in a population of ALS patients using multidimensional biomarkers. The main questions it aims to answer are:

* Which set of biomarkers explain genotypic-phenotypic correlations in ALS?
* Which set of biomarkers can be used to subdivide the ALS population in homogeneous subgroups?

Participants will undergo:

* neurological evaluation
* neurophysiological evaluation
* neuropsychological evaluation
* whole exome sequencing
* biomarker measurement in CSF and plasma

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ALS or other motor neuron disease
* residence near the study centers

Exclusion Criteria:

* refusal to participate to the study
* unable/unwilling to perform follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cohort of incident patients from three Italian ALS Centers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
genetic screening | baseline (at diagnosis)
  no. of patients with ALS-associated mutations
biomarker assessment | baseline (at diagnosis), at 6 months, at 1 year
  no. of patients with abnormal NfL, GFAP, tau, UCHL1, MCP1 and TDP-43 levels

SECONDARY OUTCOMES:
clinical assessment | baseline (at diagnosis), at 6 months, at 1 year
  no. of patients with increasing vs decreasing PUMNS/LMNS scores
neuropsychological assessment | baseline (at diagnosis), at 1 year
  no. of patients with increasing vs decreasing ECAS scores

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale San Raffaele, Milan, MI
  - Ospedale San Luca, Milan, MI
  - AOU Città della Salute e della Scienza, Torino, TO